CLINICAL TRIAL: NCT02791867
Title: Comparison of Laboratory Changes, Food Intake and Metabolic Profile in Patients With Obesity and Type2 Diabetes Mellitus: Before, During and After Taking AphoelineBrake
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study drug was not provided resulting in termination for unacceptable delays
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: RA 2014-019
Record Dates: First submitted 2016-05-12; First posted 2016-06-07 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Active (Active Comparator): AphoelineBrake administration
  Interventions: Drug: AphoelineBrake
- Placebo (Placebo Comparator): Placebo Administration
  Interventions: Drug: AphoelineBrake

INTERVENTIONS:
Drug: AphoelineBrake — The study is proposed as a placebo controlled randomized controlled trial with an intervention (AphoelineBrake) in addition to their standard treatment in comparison to a standard treatment control arm receiving an identical placebo. Prior to the commencement of any study procedures, participants will document informed consent and acknowledgement of privacy rights. Participants will be seen for initial consenting procedures, initial study procedures, and follow-up procedures at the Dasman Diabetes Institute clinic.Scheduled study visits will occur at Day 0, Day 7, Months: 1, 3, 6, 9, and 12 months in accordance with standards of medical care.

SUMMARY:
The primary objective is to determine if subjects taking the natural product AphoelineBrake™ in addition to their standard treatment experience differences in metabolic disease control, gastrointestinal hormones and inflammatory markers diet, hunger, satiety, weight, compared to patients taking a placebo in addition to their standard treatment. The secondary objective is to study the effect of Aphoeline Brake on oxidative and inflammatory stress markers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Diagnosis of T2DM
* Metformin as first line treatment
* HbA1c ≥7
* Calculated HOMA-IR ≥3.0,
* BMI 25-45
* Triglyceride level ≥ 2.26 mmol/L

Exclusion Criteria:

* Age <21 years of age
* BMI ≤ 25
* Pregnant
* Subjects on chronic nonsteroidal anti-inflammatory drugs or systemic corticosteroids.
* Subjects treated with Liraglutide (Victoza®).
* Renal, hepatic or cardiac failure.
* Subjects with a significant clinical illness within a month before the first administration of Aphoeline Brake™
* Subjects diagnosed with Irritable Bowel Syndrome.
* Subjects diagnosed with Ulcerative Colitis or Crohn's disease.
* History of significant gastrointestinal disease.
* Poor venous access.
* Poor likelihood to adhere with study procedures, as documented during the MyFitnessPal procedures prior to use of Aphoeline Brake™

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Reduction in Insulin Resistance measured by HOMA-IR | 12 months from intervention
  Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin levels.
Reduction in glycated Haemoglobin measured: HBA1c | 12 months from intervention
  HbA1c refers to glycated haemoglobin. It develops when haemoglobin, joins with glucose in the blood.

SECONDARY OUTCOMES:
Reduction in serum triglyceride level (mmol/l) | 12 months from intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Zghoul, PhD, Principal Investigator — Dasman Diabetes Institute; Jerome Schentag, PharmD, Principal Investigator — University at Buffalo, New York
Locations (1):
- Dasman DIabetes Institute, Kuwait City, Kuwait